CLINICAL TRIAL: NCT02045368
Title: STM-02: Phase I Study of IGF-Methotrexate Conjugate in the Treatment of Advanced Tumors Expressing Insulin-like Growth Factor Receptor 1 (IGF-1R)
Brief Title: Study of Insulin-like Growth Factor (IGF)-Methotrexate Conjugate in the Treatment of Advanced Tumors Expressing IGF-1R
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: IGF Oncology, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STM-02; 2013-0655 (Other: University of Illinois at Chicago (UIC) Office for the Protection of Research Subjects (OPRS))
Record Dates: First submitted 2014-01-15; First posted 2014-01-24 (Estimated); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer; Brain Cancer; Gastrointestinal Cancers; Genitourinary Cancers; Gynecologic Cancers; Head and Neck Cancers; Melanoma; Thoracic Cancers
Keywords: refractory; intolerant; solid tumors
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms; Gastrointestinal Neoplasms; Urogenital Neoplasms; Head and Neck Neoplasms; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Subject Treatment with IGF-Methotrexate conjugate (Experimental): IV infusion at the assigned dose administered on days 1, 8, and 15 of a 28 day (4 week) cycle.
  Interventions: Drug: IGF-Methotrexate conjugate

INTERVENTIONS:
Drug: IGF-Methotrexate conjugate — IV infusion at the assigned dose administered on days 1, 8, and 15 of a 28 day (4 week) cycle. Up to 7 dose levels will be tested, starting with 0.05 microequivalents per kg and up to 2.5 microequivalents per kg.
  Other Names: 765IGF-MTX

SUMMARY:
This phase I dose escalation study will evaluate IGF-Methotrexate conjugate (765IGF-MTX) in patients with advanced, previously treated tumors. 765IGF-MTX is administered as an IV infusion over 1 hour on days 1, 8 and 15 of a 28 day cycle. Treatment continues until disease progression, unacceptable toxicity, or patient refusal. Assessment of response will be confirmed with imaging studies performed at the end of cycle 2 +/- 7 days, and every 2 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of advanced malignancy, refractory to or intolerant to standard therapy and is no longer likely to respond to such therapy.
2. Tumor (tissue, bone marrow, or blood) must express IGF-1R, defined as 10% or higher of cells expressing IGF-1R by immuno-histochemistry (IHC), or 0.1% or higher for IGF-1R expression by flow cytometry (blood or bone marrow aspirate).
3. Paraffin-embedded tissue sections will be stained with antibodies against insulin-like growth factor receptor 1 (IGFR-1) according to the manufacturer's recommended protocols. IHC staining and flow cytometry will be performed at the Pathology Department of the University of Illinois Cancer Center.
4. Measurable or evaluable disease per RECIST 1.1 criteria for solid tumors and lymphoma as defined in the protocol. For other hematologic malignancies, see below (measurable disease per RECIST 1.1 criteria not necessary).
5. Multiple Myeloma: Confirmed diagnosis of multiple myeloma as defined in the protocol with relapsed or refractory disease, and measurable disease defined as one of below:

   * Serum monoclonal protein > 500mg/dL by serum protein electrophoresis (SPEP)
   * Urine monoclonal protein > 200mg/24 hours by urine protein electrophoresis (UPEP)
   * Measurable free light chain by free light chain assay > 10mg/dL with abnormal kappa to lambda light chain ratio
   * Measurable bone disease by > 1 bone lesion which is > 20 mm on conventional techniques or > 10 mm with spiral CT (for lytic lesions)
   * Monoclonal bone marrow plasmacytosis > 30%
6. Lymphoma: Previously treated, histologically confirmed lymphoma with measurable disease via RECIST 1.1, with the exception of lymphoplasmacytic lymphoma, which can be diagnosed based on morphologic evidence in the bone marrow plus the appropriate paraprotein.
7. Waldenstrom's Macroglobulinemia: Confirmed diagnosis with relapsed or refractory disease, and measurable disease defined as at least one lesion with a single diameter of greater than 2cm by CT or bone marrow involvement with greater than 10% malignant cells and immunoglobulin (IgM, IgG, IgA) greater than 1000mg/dL.
8. Hematologic malignancies including myelodysplastic syndrome(MDS), leukemia: Confirmed histologic diagnosis with relapsed or refractory disease; measurable disease per RECIST 1.1 criteria is not required.
9. Age ≥ 18 years
10. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
11. Prior systemic chemotherapy, immunotherapy, or biological therapy, radiation therapy and/or surgery are allowed; however prior use of methotrexate allowed if > 6 months prior to study entry. Intrathecal methotrexate is allowed prior to and during treatment per investigator discretion. Time since prior therapy and the first dose of study drug:

    * At least 2 weeks since prior radiation, non cytotoxic small molecule drugs (e.g., tyrosine kinase inhibitors such as erlotinib and hormonal agents such as letrozole), prior major surgery (surgery defined as a surgery involving a risk to the life of the patient; specifically: an operation upon an organ within the cranium, chest, abdomen, or pelvic cavity), prior systemic FDA approved therapy

      * At least 3 weeks since prior antineoplastic therapy
      * At least 4 weeks since exposure to monoclonal antibodies (chimeric or fully human)
      * At least 6 weeks since prior nitrosureas or mitomycin-C
12. Patient must have recovered from the acute toxic effects (≤ grade 1 CTCAE v.4.0) of previous anti-cancer treatment prior to study enrollment; the only exception is that grade 2 neuropathy is permitted
13. Adequate organ function within 14 days of study registration defined as the following laboratory values:

    * Absolute neutrophil count (ANC) ≥ 1.5 X 10^9/L
    * Hemoglobin ≥ 9g/dL* (Patient may not have had a transfusion within 7 days of blood draw.)
    * Platelets ≥ 100 X 10^9/L* (Patient may not have had a transfusion within 7 days of blood draw.)
    * Total bilirubin ≤ 1.5 X upper limit of normal (ULN)
    * Alkaline phosphatase, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 X ULN < 5 X ULN is acceptable if liver has tumor involvement)
    * Serum creatinine ≤ 1.5 X ULN
    * Creatinine clearance ≥ 60 ml/min^2 or glomerular filtration rate (GFR) ≥ 60 ml/min^2 or 24 hour urine creatinine clearance ≥ 50 ml/min
    * Laboratory values for lymphoma patients:

      * Absolute neutrophil count (ANC) ≥ 1.0 X 10^9/L
      * Hemoglobin ≥ 8g/dL
      * Platelets ≥ 50 X 10^9/L
      * Total bilirubin ≤ 1.5 X ULN
      * Alkaline phosphatase, AST and ALT ≤ 3 X ULN (< 5 X ULN is acceptable if liver has tumor involvement)
      * Serum creatinine ≤ 1.5 X ULN
      * Creatinine clearance ≥ 60 ml/min^2 or GFR ≥ 60 ml/min^2 or 24 hour urine creatinine clearance ≥ 50 ml/min
14. Negative urine or serum pregnancy test in females. Male and female patients with reproductive potential must use an approved contraceptive method if appropriate (for example, abstinence, oral contraceptives, implantable hormonal contraceptives, or double barrier methods) during and for 3 months after the last dose of 765IGF-MTX.
15. Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.

Exclusion Criteria:

1. Untreated central nervous system (CNS) metastases
2. Radiation therapy to more than 25% of the bone marrow. Whole pelvic radiation is considered to be over 25%.
3. ≥ Grade 3 peripheral neuropathy within 14 days before enrollment.
4. Systemic infection requiring IV antibiotic therapy within 7 days preceding the first dose of study drug, or other severe infection.
5. Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
6. Pregnant or breastfeeding - methotrexate is Pregnancy Category X - has been reported to cause fetal death and/or congenital abnormalities. Confirmation that the subject is not pregnant must be established by a negative serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
7. Uncontrolled diabetes mellitus defined as a Hemoglobin A1C≥ 7% in patients with a prior history of diabetes, 28 days prior to study enrollment.
8. Serious concomitant systemic disorders (e.g., active infection, uncontrolled diabetes) or psychiatric disorders that, in the opinion of the investigator, would compromise the safety of the patient or compromise the patient's ability to complete the study.
9. Other severe acute or chronic medical or psychiatric conditions, or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for enrollment in this study.
10. Recent (within 6 months) arterial thromboembolic events, including transient ischemic attack (TIA), cerebrovascular accident (CVA), unstable angina, or myocardial infarction (MI).
11. History of abdominal fistula, gastrointestinal perforation, or intra abdominal abscess within 28 days prior to beginning study treatment.
12. Abnormalities on 12-lead electrocardiogram (ECG) considered by the investigator to be clinical significant.
13. History of cerebrovascular accident, pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months. Note: Subjects with recent DVT who have been treated with therapeutic anticoagulants for at least 6 weeks are eligible.
14. Presence of any non-healing wound, fracture, or ulcer within 28 days prior to the first dose of study drug.
15. Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to IGF or methotrexate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2014-01-28 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Up to 30 days after final dose.
  The primary objective is to determine the maximum tolerated dose (MTD) of 765IGF-MTX by evaluation of toxicity for the treatment of advanced, previously treated malignancies that express IGF-1R.

SECONDARY OUTCOMES:
Adverse Effects | Up to 30 days after last dose study drug.
  Characterize adverse effects (AE) of 765IGF-MTX in patients with advanced, previously treated malignancies as defined by CTCAE v 4.0.
Disease Response based on RECIST Criteria | Up to 8 weeks after last dose study drug.
  Evaluate clinical response of 765IGF-MTX in patients with advanced, previously treated malignancies. Disease response will be assessed every 8 weeks while on study treatment using the Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST 1.1).

CONTACTS AND LOCATIONS:
Overall Officials: Neeta Venepalli, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No